CLINICAL TRIAL: NCT00850356
Title: Alberta Population-based, Prospective Evaluation of the Quality of Life Outcomes and Economic Impacts of Bariatric Surgery
Brief Title: Quality of Life Outcomes and Economic Impacts of Bariatric Surgery
Status: Completed | Type: Observational
Sponsor: University of Alberta (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Raj Padwal, Associate Professor, General Internal Medicine, University of Alberta
Other Study IDs: #B-120208
Record Dates: First submitted 2009-02-24; First posted 2009-02-25 (Estimated); Last update posted 2013-05-21 (Estimated); Status verified 2013-05

CONDITIONS: Obesity
Keywords: Bariatric Surgery; Body Weight; Health care costs; Obesity; Obesity Complications; Prolonged wait times; Quality of Life
MeSH Terms: conditions — Obesity; Body Weight

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (3):
- Bariatric Surgery Patient (Sx): Participants who are patients in an Adult Weight Management Clinic (AWMC) and undergo bariatric surgery.
- Medical Treamtent (Mx): Participants who are patients in the same AWMC as above and are currently undergoing a medical treatment program that includes intensive lifestyle counseling (diets, exercise, behavioral modification).
- Wait-List (Wx): Participants who are on the Wait-List for the AWMC, and waiting to undergo medical treatment program and/or bariatric surgery.

SUMMARY:
The purpose is to determine the economic, clinical and quality of life outcomes of bariatric surgery and describe the consequences of protracted wait-times (~ 2 years) for this procedure.

DETAILED DESCRIPTION:
Severe obesity affects approximately 3% of Canadians (nearly 1 million people) and is becoming increasingly common and costly. Surgery for severe obesity, known as bariatric surgery, substantially reduces weight and the risk of death, decreases obesity-related health problems and increases quality of life. However, surgery carries a 0.5-2% up-front risk of death, has potentially serious short and long-term complications, and an uncertain cost-to-benefit ratio. Surgery is becoming increasingly popular, programs are being initiated or expanded across the country, and waiting lists are several years long. Provincial governments, unable to keep pace with surgical demand, are sending patients to the US for surgery and patients are petitioning governments for increased access to care.

By collecting data from a clinical obesity program that services an entire Canadian health region of over 1 million people and linking these data to provincial and regional data sources, this study aims to:

1. Determine whether surgery improves 2-yr medical and patient-centered outcomes (such as quality of life, satisfaction, and others) compared to both medical and community wait-list control patients;
2. Comprehensively compare the 3-yr costs of surgical and non-surgical care;
3. Determine the impact of 2-yr wait times for surgery on patient health and wellness, including quality of life and patient satisfaction.

This study will provide essential data to accurately determine the benefits, risks, and costs of bariatric surgery in the Canadian context for patients, care providers, and decision makers. Equally important, it will determine whether the health and quality of life of Canadians waiting for surgery is adversely affected because of extended wait-times. Results will directly influence and streamline patient care, will be applicable to similar programs across the country, and serve as an important foundation for future research and data collection.

ELIGIBILITY:
Inclusion Criteria:

1. 18-60 years old
2. Male and Female
3. BMI Levels greater than or equal to 35 kg/m2 and a major medical comorbidity OR BMI levels greater than or equal to 40 kg/m2
4. Able to provide written informed consent

Exclusion Criteria:

1. Pregnant or nursing
2. Previously enrolled in this study (e.g Community Control Arm)
3. Currently participating in a clinical trial
4. Individual expected to have difficulty with follow-up visits, completion of questionnaires, etc.
5. Any contraindications to bariatric surgery and/or anti-obesity medical treatment
6. Ability and willingness to complete questionnaires.
7. Any other medical, social or geographic condition, which, in the opinion of the investigator would not allow safe completion of the study protocol.
8. Patients in whom protein sparing very low calorie diet therapy is planned.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Three participant goups (n=500:)
  Bariatric Surgery(Sx):150 participants. Patients approved for bariatric surgery in an Adult Weight Management Clinic (AWMC) will be eligible (BMI ≥35 kg/m2 and a major medical comorbidity or BMI ≥ 40 kg/m2). Contraindications to surgery are pregnancy, unstable psychiatric disease, patients deemed too medically high-risk, age > 60 years, active substance abuse, or an active eating disorder.
  Medical Treatment(Mx):200 participants. Patients will be approached for the study upon their first visit in the AWMC.
  Both medical and surgical patients receive intensive lifestyle counseling (diets, exercise, behavioral modification) delivered according to current recommendations. Other than receiving extra education about surgery and post-operative diets, there is no difference in care between the medical and surgical arms.
  Community Wait-List Control(Wx):150 participants will be enrolled from the list of newly referred patients to the AWMC.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2008-11; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Quality of life measured through responses to standardized health questionnaires: SF-12; EQ-5D; IWQoL(Impact of Weight on Quality of Life); PSS(Patient satisfaction survey); Mod WLIQ:(Modified Waiting-list impact questionnaire) | Every Six months for 2 years (At time =0, 6, 12, 18, 24 months)

SECONDARY OUTCOMES:
Comprehensive comparison of the 3-yr costs of surgical and non-surgical care through medication logs, a questionnaire package, and accessing Alberta health and Wellness data. | Every six months for 2 years (At time =0, 6, 12, 18, 24 months)

CONTACTS AND LOCATIONS:
Overall Officials: Raj Padwal, MD, Principal Investigator — University of Alberta
Locations (1):
- Royal Alexandra Hospital, Edmonton, Alberta, Canada

REFERENCES:
- [Background] Padwal RS, Chang HJ, Klarenbach S, Sharma AM, Majumdar SR. Characteristics of the population eligible for and receiving publicly funded bariatric surgery in Canada. Int J Equity Health. 2012 Sep 18;11:54. doi: 10.1186/1475-9276-11-54. PMID 22984790
- [Background] Padwal RS, Majumdar SR, Klarenbach S, Birch DW, Karmali S, McCargar L, Fassbender K, Sharma AM. The Alberta population-based prospective evaluation of the quality of life outcomes and economic impact of bariatric surgery (APPLES) study: background, design and rationale. BMC Health Serv Res. 2010 Oct 8;10:284. doi: 10.1186/1472-6963-10-284. PMID 20932316
- [Result] Padwal RS, Majumdar SR, Klarenbach S, Birch DW, Karmali S, McCargar L, Fassbender K, Sharma AM. Health status, quality of life, and satisfaction of patients awaiting multidisciplinary bariatric care. BMC Health Serv Res. 2012 Jun 8;12:139. doi: 10.1186/1472-6963-12-139. PMID 22681857
- [Derived] Warkentin LM, Majumdar SR, Johnson JA, Agborsangaya CB, Rueda-Clausen CF, Sharma AM, Klarenbach SW, Karmali S, Birch DW, Padwal RS. Weight loss required by the severely obese to achieve clinically important differences in health-related quality of life: two-year prospective cohort study. BMC Med. 2014 Oct 15;12:175. doi: 10.1186/s12916-014-0175-5. PMID 25315502
- [Derived] Padwal RS, Rueda-Clausen CF, Sharma AM, Agborsangaya CB, Klarenbach S, Birch DW, Karmali S, McCargar L, Majumdar SR. Weight loss and outcomes in wait-listed, medically managed, and surgically treated patients enrolled in a population-based Bariatric program: prospective cohort study. Med Care. 2014 Mar;52(3):208-15. doi: 10.1097/MLR.0000000000000070. PMID 24374423